CLINICAL TRIAL: NCT02655809
Title: Physica KR: In Vivo Kinematic Analysis of a Novel Total Knee Replacement Implant
Brief Title: Physica KR Fluoroscopy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Limacorporate S.p.a (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: K-07
Record Dates: First submitted 2016-01-08; First posted 2016-01-14 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Total Knee Replacement

ARMS (1):
- Physica KR (Other): Patients who have received a Physica KR total knee implant.
  Interventions: Radiation: Fluoroscopic examination

INTERVENTIONS:
Radiation: Fluoroscopic examination

SUMMARY:
The aim of this study is to assess the in vivo kinematics and range of motion of a single-surgeon clinical series of TKA performed with a fixed-bearing cruciate retaining total knee arthroplasty that has a roll-back mechanism and compare it with the kinematic of the normal healthy knee.

Patients would be evaluated by fluoroscopic examination during weight bearing activities (lounging, kneeling and stairs climbing).

ELIGIBILITY:
Inclusion Criteria:

1. Patientsoperated in The Royal Bournemouth Hospital NHS Foundation Trust and who has received a Physica KR implant
2. Patients achieving a ROM ≥ 100° at 6 week follow-up in the Physica KR clinical trial (K-06 Study protocol 30/10/2013 v 1.0);
3. Patients affected by primary or secondary OA before surgery;
4. Patients with an appropriate intial fixation and stability of the knee prosthesis;
5. Patients with undamaged and functional collateral and posterior cruciate ligaments (no ligamentous imbalance or pain);
6. Patients who understand the requirements of the study and are willing and able to comply with activities required for fluoroscopic examination;
7. Patients who have signed the Ethics Committee approved study-specific Informed Consent Form.

Exclusion Criteria:

1. Patients with a ROM < 100° at 6-week follow-up in Physica KR clinical trial (K-06- Study protocol 30/10/2013 v 1.0);
2. Patients affected by rheumatoid arthritis;
3. Patients with malalignment or axial malrotation of the knee prosthesis;
4. Patients who had or have planned a surgery on their uninvolved knee within a year;
5. Muscular insufficiency or absence of muscoligamentous supporting structures required for adequate soft tissue balance;
6. Patients who have significant neurological or musculoskeletal disorders or disease that may adversely affect gait and compromise functional recovery and evaluation;
7. Patients who have neuromuscular or neurosensory deficit which would limit the ability to assess the performance of the device;
8. Any psychiatric illness that would prevent comprehension of the details and nature of the study;
9. Participation in any experimental drug/device study within the 6 months prior to the preoperative visit, excluding the Physica KR clinical trial (K-06 Study protocol 30/10/2013 v 1.0);
10. Female patients who are pregnant, nursing, or planning a pregnancy.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Assessment of the roll-back mechanism by measuring the contact point between tibia and femur components in millimeters | 6 months after surgery
  Using a software to replicate the movement using CAD models. The movement is studied and the distance made by the femur on the tibia is calculated giving the information of the roll back.

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Bournemouth Hospital, Bournemouth, Dorset, United Kingdom